CLINICAL TRIAL: NCT01048203
Title: An Open Label, Single Dose Metabolism and Mass Balance Study of 14C-ABR-215050 in Healthy Subjects
Brief Title: A Single Dose Metabolism and Mass Balance Study of 14C-ABR-215050 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Active Biotech AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 08TASQ09; 2008-003163-39 (EudraCT Number)
Record Dates: First submitted 2010-01-08; First posted 2010-01-13 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
Keywords: 14C ABR 215050 Metabolism and Mass Balance Study; tasquinimod; Metabolic pattern of 14C ABR-215050
MeSH Terms: interventions — tasquinimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ABR-215050 (Experimental)
  Interventions: Drug: ABR-215050

INTERVENTIONS:
Drug: ABR-215050 — 1 mg ABR-215050
  Other Names: tasquinimod

SUMMARY:
This is a single site, open label, single dose, non-randomized study in healthy male and female subjects. The subjects will be evaluated for plasma, urine and feces levels of 14C-ABR-215050 during 21 days.

DETAILED DESCRIPTION:
As a part of the pharmacokinetic documentation, the metabolism and mass balance of 14C-ABR-215050 will be studied in healthy subjects. Female healthy subjects are included in the study in case of expanding the indication to female forms of cancer. In this study a single dose of 1.0 mg of the study drug will be administered orally as a solution under fasted conditions. The absorption and safety profiles for the oral water solution will also be documented.

ELIGIBILITY:
Inclusion Criteria:

1. 40-65 year old male and female subjects.
2. Healthy according to medical history, physical examination and clinical chemistry, urine and hematological laboratory tests.
3. Body Mass Index (BMI) of 18-30.
4. Negative screen for Hepatitis B / C and HIV-infection.
5. Be willing and able to comply with the protocol for the duration of the study.
6. Women of childbearing potential must be neither pregnant nor breast-feeding. Confirmation that the subject is not pregnant must be established by a pregnancy test before the single dose and at study end. Fertile women must be willing to practice reliable methods of contraception. Medically accepted safe methods of contraception for the purpose of this study will include surgical sterilisation, intra-uterine device, diaphragm with spermicide, or condom with spermicide. As interaction studies between ABR-215050 and hormonal (oral or depot) contraceptives have not yet been performed, women using such devices must also use a complementary contraceptive device.
7. Have given written signed informed consent, prior to start of any study-related activities.

Exclusion Criteria:

1. Gastrointestinal disorders that may affect drug absorption.
2. Any vaccination within 30 days before start of this study and throughout the study.
3. Blood donation within 90 days before start of this study and for 90 days after the study.
4. Participation in other clinical studies or who have received other investigational drugs within 90 days prior to enrolment. Additionally, subjects previously included into this study and then are withdrawn from the study is not to be re-entered into the study.
5. Perform any planned surgery
6. Any use of nicotine within three (3) months before start of this study and throughout the study.
7. Known or suspected history of alcoholism or drug abuse.
8. Intake of alcoholic beverages for 24 hours prior to the administration of investigational product and for 24 hours after the dose.
9. Intake of caffeine containing beverages 10 hours prior to the administration of investigational product and for 6 hours after the dose.
10. Medication including herbal remedies (vitamins and paracetamol excluded) within 14 days before and throughout the study.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To establish the metabolic pattern of ABR 215050 | 4 months

SECONDARY OUTCOMES:
To study the mass balance and to determine the disposition and pathways of elimination of 14C-ABR-215050. | 4 months
To follow the safety profile | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Ellman, BSc, Study Director — Active Biotech Research AB
Locations (1):
- JJ Berzelius Clinical Research Center AB, Berzelius Science Park, Linköping, Sweden